CLINICAL TRIAL: NCT01814800
Title: An Open Label, Multicenter, Study to Evaluate the Pharmacokinetics, Efficacy and Safety of RI-002 (IGIV) in Subjects With Primary Immunodeficiency Diseases (PIDD)
Brief Title: Pharmacokinetics, Efficacy, and Safety Study of RI-002 (IGIV) in Subjects With Primary Immunodeficiency Diseases (PIDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADMA-003
Record Dates: First submitted 2013-03-06; First posted 2013-03-20 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: PIDD, PID, humoral immunity, antibody deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RI-002 Treatment (Experimental): Drug: RI-002 Dose: 300-800 mg/kg infusion Frequency: Once every 3 to 4 Weeks
  Interventions: Biological: RI-002

INTERVENTIONS:
Biological: RI-002 — Immune Globulin Intravenous (IGIV)
  Other Names: Immune Globulin (Human)

SUMMARY:
This is a Phase III, multicenter, open-label study of RI-002 administered as an intravenous infusion of RI-002 (IGIV) every 21 or 28 days in approximately 60 subjects with Primary Immunodeficiency Diseases (PIDD).

DETAILED DESCRIPTION:
Primary immunodeficiency diseases (PIDDs) are genetically determined disorders of the immune system resulting in greatly enhanced susceptibility to infectious disease, autoimmunity and malignancy. As most subjects with PIDDs present with infections, the differential diagnosis and initial investigations for an underlying immune defect are typically guided by the clinical presentation. In subjects with PIDDs, individual infections are not necessarily more severe than those that occur in a normal host. Rather, the clinical features suggestive of an immune defect may be the recurring and/or chronic nature of infections with common pathogens that may result in end organ damage, such as bronchiectasis. Several immune globulin products have already been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, the subjects must meet the following criteria:

1. Signed a written informed consent or a specific assent form for minors.
2. Have a diagnosis of primary immunodeficiency disease.
3. Be ≥ 2 years and ≤ 75 years.
4. Have body weight ≥ 12 kg at screening.
5. Have been receiving IGIV at a dose that has not been changed by >50% of the mean dose on a mg/kg basis for at least 3 months prior to study entry and have maintained a trough serum Immunoglobulin G (IgG) level ≥ 500 mg/dL on the previous 2 assessments prior to receiving RI 002. The trough level must be at least 300 mg/dL above the pre-treatment serum IgG level.
6. For female subjects, be of non-childbearing potential or have a negative pregnancy test prior to study start and be deemed not at risk of becoming pregnant by adherence to a reliable contraceptive method for the duration of the study.

Exclusion Criteria:

Subjects must be excluded if they meet any of the following criteria:

1. Have a known hypersensitivity to immunoglobulin or any excipient in RI-002.
2. Have a history of a severe anaphylactic or anaphylactoid reaction to blood or any blood-derived product.
3. Have a specific Immunoglobulin A (IgA) deficiency, history of allergic reaction to products containing IgA or has demonstrable antibodies to IgA.
4. Have uncompensated hemodynamically significant congenital or other heart disease.
5. Have a medical condition that is known to cause secondary immune deficiency.
6. Have a significant T-cell deficiency or deficiency of granulocyte number or function.
7. Have significant renal impairment or have a history of acute renal failure.
8. Have abnormal liver function.
9. Be receiving chronic anti-coagulation therapy.
10. Have a history of deep vein thrombosis (DVT), thrombotic or thrombo-embolic event, or are at increased risk for thrombotic events.
11. Current daily use of the following medications:

    * corticosteroids (> 7.5 mg (or equivalent dose on a mg/kg basis) of prednisone equivalent per day for > 30 days)
    * immunomodulatory drugs
    * immunosuppressive drugs (excluding topical pimecrolimus (Elidel) and tacrolimus (Protopic))
12. Administration of a hyperimmune or specialty high titer immunoglobulin product.
13. Have uncontrollable arterial hypertension.
14. Have a history of hemolysis or positive Coombs test while undergoing treatment with IGIV therapy.
15. Be morbidly obese as indicated by a Body Mass Index (BMI) ≥ 40
16. Have received any blood product (other than Immunoglobulin G) within 3 months prior to screening.
17. Have received any Respiratory Syncytial Virus (RSV) specific products, including palivizumab (Synagis®) within 3 months prior to screening.
18. Have abused alcohol, opiates, psychotropic agents, or other chemicals or drugs within the past 12 months.
19. Have any condition or abnormal laboratory assessment judged by the investigator to preclude participation in the study.
20. Are currently pregnant or nursing.
21. Have hepatitis A, B, or C.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Mond, M.D., Ph.D., Study Director — ADMA Biologics, Inc.
Locations (9):
- United States (9):
  - IMMUNOe Health Centers, Cenntennial, Colorado
  - Allergy Associates of the Palm Beaches, P.A., North Palm Beach, Florida
  - Family Allergy Center, PC, Atlanta, Georgia
  - The South Bend Clinic, LLP, South Bend, Indiana
  - Asthma & Immunology Associates, Omaha, Nebraska
  - Mount Sinai School of Medicine, New York, New York
  - Dallas Immunology Research, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - Baylor Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- RI-002 Treatment: Drug: RI-002 Dose: 300-800 mg/kg IV infusion Frequency: Every 3 or 4 weeks
  Initial dose selection based on prior IGIV regimen, doses adjusted during study to maintain trough Immunoglobulin G (IgG) concentration of 500 mg/dL or greater according to investigator decision.
Period: Overall Study
Arm/Group | RI-002 Treatment
Started | 59
Completed | 54
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Pregnancy | 1
Not completed — Sponsor decision | 1
Not completed — Subject relocation | 1

BASELINE CHARACTERISTICS:
Groups:
- RI-002 Treatment: Drug: RI-002 Dose: 300-800 mg/kg infusion
  RI-002
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 35
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 41.8 [3 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 59
PIDD Type [Number; unit: participants] — Primary PIDD diagnosis
  participants
    Common Variable Immunodeficiency | 45
    X-Linked Agammaglobulinemia | 6
    Antibody Deficiencies | 4
    Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Bacterial Infections (SBIs) Per Subject Per Year (FDA Guidance for Industry (2008))
Description: The primary objective of this study was to demonstrate that RI-002 (IGIV) reduces the frequency of serious bacterial infections (SBIs), as defined by the Diagnostic Criteria for Serious Infection Types guideline, in subjects with primary humoral immunodeficiency.
Time Frame: One year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: SBIs/subject/year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
SBIs/subject/year | 0

2. Secondary Outcome: Incidence of All Infections (Serious and Non-serious)
Time Frame: Up to 1 Year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: events per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
events per subject-year
  Number of Infections (All) per subject-year | 3.436
  Number of Serious Infections per subject-year | 0.018

3. Secondary Outcome: Number of Days Lost From Work/School/Daycare and Usual Activities Due to Infections and Their Treatment - Combined Days Lost
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days | 243

4. Secondary Outcome: Number of Days Lost From Work/School/Daycare and Usual Activities Due to Infections and Their Treatment - Per Subject-Year
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days per subject-year | 4.349

5. Secondary Outcome: Number of Unscheduled Visits to Physician/ER Due to Infections - Total Number of Visits
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Number of Visits
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Number of Visits | 54

6. Secondary Outcome: Number of Unscheduled Visits to Physician/ER Due to Infections - Per Subject-Year
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Number of Visits per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Number of Visits per subject-year | 0.966

7. Secondary Outcome: Time to Resolution of Infections - Duration Per Infection
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days | 16.7 (27.83)

8. Secondary Outcome: Time to Resolution of Infections - Infection Days Per Subject
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Mean (Standard Deviation); unit: Days per subject
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days per subject | 62.7 (86.80)

9. Secondary Outcome: Number of Hospitalizations Due to Infections
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Number of hospitalizations
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Number of hospitalizations | 1

10. Secondary Outcome: Number of Hospitalizations Due to Infections - Per Subject-Year
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Hospitalizations per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Hospitalizations per subject-year | 0.018

11. Secondary Outcome: Days of Hospitalization Due to Infections
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days | 5

12. Secondary Outcome: Days of Hospitalization Due to Infections - Per Subject-Year
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days per subject-year | 0.089

13. Secondary Outcome: Number of Days of Antibiotic Therapy (Prophylaxis and Treatment of Infection)
Description: Summary of the days of antibiotic therapy in the study for prophylaxis, as treatment for infections, and combined
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days
  Total days of antibiotic use COMBINED | 2969
  Total days of antibiotic use for INFECTION | 1839
  Total days of antibiotic use for PROPHYLAXIS | 1130

14. Secondary Outcome: Number of Days of Antibiotic Therapy (Prophylaxis and Treatment of Infection) - Per Subject-Year
Description: Summary of the days of antibiotic therapy in the study for prophylaxis, as treatment for infections, and combined, per subject-year of treatment with RI-002
Time Frame: Up to 1 year
Population: Analysis included 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days per subject-year
  Days of antibiotic use per subject-year COMBINED | 53.135
  Days of antibiotic per subject-year for INFECTION | 32.912
  Days of antibiotic per subject-yr for PROPHYLAXIS | 20.223

15. Secondary Outcome: Correlation Between Trough Level of RI-002 and Serious and Non-serious Infections
Description: The relationship between trough IgG concentrations and the number of infections of any kind/seriousness was evaluated using Pearson linear correlation coefficients using forward analysis (outcomes after infusion) and backward analysis (outcomes prior to infusion; outcomes post last infusion were excluded)
Time Frame: Up to 1 year
Measure: Number; unit: Linear Correlation Coefficients
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Linear Correlation Coefficients
  Forward analysis | -0.0453
  Backward analysis | -0.0045

16. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - IgG
Description: Summary of trough total IgG concentration prior to specified infusion
Time Frame: Up to 1 year
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
mg/dL
  Infusion 1 (n=59) | 1000 (36.32)
  Infusion 2 (n=57) | 1024.3 (33.38)
  Infusion 3 (n=55) | 1007.5 (33.26)
  Infusion 4 (n=56) | 1017.4 (34.96)
  Infusion 5 (n=55) | 1008.1 (32.49)
  Infusion 6 (n=56) | 1016.1 (34.18)
  Infusion 7 (n=55) | 1039.5 (37.50)
  Infusion 8 (n=56) | 957.7 (35.49)
  Infusion 9 (n=56) | 1030.5 (36.77)
  Infusion 10 (n=54) | 1021.7 (37.27)
  Infusion 11 (n=55) | 1018.9 (34.85)
  Infusion 12 (n=54) | 1000.6 (33.62)
  Infusion 13 (n=53) | 992.8 (35.34)
  Infusion 14 (3-week cycle only) (n=16) | 1165.3 (79.59)
  Infusion 15 (3-week cycle only) (n=16) | 1160.9 (77.96)
  Infusion 16 (3-week cycle only) (n=16) | 1147.9 (74.93)
  Infusion 17 (3-week cycle only) (n=16) | 1136.3 (70.78)

17. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Haemophilus Influenzae Type B
Description: Summary of trough antibody concentrations prior to specified infusion for Haemophilus influenzae type B
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 3.25 (0.417)
  Infusion 4 (n=56) | 3.12 (0.454)
  Infusion 8 (n=56) | 2.93 (0.364)
  Infusion 12 (n=54) | 3.11 (0.442)
  End of Study (Infusion 13 / 17) (n=53) | 3.31 (0.404)

18. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Respiratory Syncytial Virus (RSV)
Description: Summary of trough antibody concentrations prior to specified infusion for Respiratory Syncytial Virus (RSV)
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 51-56 subjects
Measure: Mean (Standard Error); unit: titer
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 56
titer
  Infusion 1 (n=56) | 1211.9 (187.13)
  Infusion 4 (n=54) | 2220.1 (286.79)
  Infusion 8 (n=54) | 1936.2 (363.84)
  Infusion 12 (n=52) | 1632.4 (224.90)
  End of Study (Infusion 13 / 17) (n=51) | 1862.3 (207.94)

19. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Tetanus
Description: Summary of trough antibody concentrations prior to specified infusion for Tetanus
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
IU/mL
  Infusion 1 (n=59) | 5.98 (0.573)
  Infusion 4 (n=56) | 7.57 (0.586)
  Infusion 8 (n=56) | 7.07 (0.523)
  Infusion 12 (n=54) | 6.97 (0.470)
  End of Study (Infusion 13 / 17) (n=53) | 6.50 (0.531)

20. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 1
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 1
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 3.108 (0.5967)
  Infusion 4 (n=55) | 2.900 (0.4585)
  Infusion 8 (n=56) | 2.866 (0.5154)
  Infusion 12 (n=54) | 2.788 (0.6185)
  End of Study (Infusion 13 / 17) (n=53) | 2.736 (0.5030)

21. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 3
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 3
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 1.447 (0.1077)
  Infusion 4 (n=56) | 1.873 (0.1263)
  Infusion 8 (n=56) | 1.787 (0.1105)
  Infusion 12 (n=54) | 1.686 (0.1360)
  End of Study (Infusion 13 / 17) (n=53) | 1.672 (0.1249)

22. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 4
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 4
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-58 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=58) | 0.530 (0.0713)
  Infusion 4 (n=56) | 0.824 (0.1589)
  Infusion 8 (n=55) | 0.610 (0.0624)
  Infusion 12 (n=53) | 0.644 (0.0703)
  End of Study (Infusion 13 / 17) (n=53) | 0.802 (0.1681)

23. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 5
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 5
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 52-58 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=58) | 10.843 (0.7116)
  Infusion 4 (n=54) | 12.264 (0.8885)
  Infusion 8 (n=55) | 11.235 (0.8974)
  Infusion 12 (n=54) | 11.707 (0.8858)
  End of Study (Infusion 13 / 17) (n=52) | 10.503 (0.8420)

24. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 6B
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 6B
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 2.121 (0.2529)
  Infusion 4 (n=56) | 2.496 (0.2503)
  Infusion 8 (n=56) | 2.166 (0.1849)
  Infusion 12 (n=54) | 2.026 (0.2199)
  End of Study (Infusion 13 / 17) (n=53) | 1.862 (0.2054)

25. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 7F
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 7F
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-57 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=57) | 3.413 (0.4009)
  Infusion 4 (n=55) | 3.457 (0.3930)
  Infusion 8 (n=55) | 2.633 (0.1971)
  Infusion 12 (n=54) | 2.492 (0.2703)
  End of Study (Infusion 13 / 17) (n=53) | 3.191 (0.4040)

26. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 9V
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 9V
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 1.473 (0.1063)
  Infusion 4 (n=56) | 1.938 (0.1566)
  Infusion 8 (n=56) | 2.010 (0.2842)
  Infusion 12 (n=53) | 1.902 (0.1579)
  End of Study (Infusion 13 / 17) (n=53) | 2.223 (0.3123)

27. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 14
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 14
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 4.853 (0.4724)
  Infusion 4 (n=56) | 6.744 (0.3984)
  Infusion 8 (n=56) | 6.356 (0.3547)
  Infusion 12 (n=54) | 6.341 (0.4275)
  End of Study (Infusion 13 / 17) (n=53) | 6.218 (0.4268)

28. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 18C
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 18C
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 7.259 (0.7462)
  Infusion 4 (n=56) | 7.461 (0.6143)
  Infusion 8 (n=55) | 6.588 (0.5627)
  Infusion 12 (n=54) | 7.146 (0.7852)
  End of Study (Infusion 13 / 17) (n=53) | 6.566 (0.5452)

29. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 19A
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 19A
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 51-54 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=53) | 19.090 (1.6428)
  Infusion 4 (n=52) | 17.717 (1.3715)
  Infusion 8 (n=54) | 15.450 (1.2636)
  Infusion 12 (n=51) | 11.621 (1.0681)
  End of Study (Infusion 13 / 17) (n=52) | 12.167 (1.4398)

30. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 19F
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 19F
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 6.630 (1.0784)
  Infusion 4 (n=55) | 7.876 (0.8826)
  Infusion 8 (n=56) | 7.361 (0.8704)
  Infusion 12 (n=53) | 7.042 (0.7610)
  End of Study (Infusion 13 / 17) (n=53) | 7.681 (0.9497)

31. Secondary Outcome: Trough Total IgG and Specific Antibody Levels - Streptococcus Pneumoniae, Serotype 23F
Description: Summary of trough antibody concentrations prior to specified infusion for Streptococcus Pneumoniae, Serotype 23F
Time Frame: Up to 1 year
Population: Number available for analysis varied by infusion; 53-59 subjects
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
ug/mL
  Infusion 1 (n=59) | 1.490 (0.1453)
  Infusion 4 (n=55) | 1.829 (0.1548)
  Infusion 8 (n=56) | 1.580 (0.1128)
  Infusion 12 (n=54) | 1.554 (0.1179)
  End of Study (Infusion 13 / 17) (n=53) | 1.681 (0.1282)

32. Post Hoc Outcome: Number of Days Lost From Work/School/Daycare Due to Infections and Their Treatment
Description: Additional analysis performed to separate the number of days lost from work, school and/or daycare from the days missed from normal activities, due to infection
Time Frame: Up to 1 year
Population: Analysis includes 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days | 93

33. Post Hoc Outcome: Number of Days Lost From Work/School/Daycare Due to Infections and Their Treatment - Per Subject-Year
Description: as for outcome 32
Time Frame: Up to 1 year
Population: Analysis includes 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: Days per subject-year
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
Days per subject-year | 1.66

34. Post Hoc Outcome: Number of Participants With No Days Lost From Work/School/Daycare Due to Infections and Their Treatment
Description: Additional analysis performed to separate the number of days lost from work, school and/or daycare from the days missed from normal activities, due to infection. Presenting the number of subjects with no (0) days lost from work/school/daycare due to infection
Time Frame: Up to 1 year
Population: Analysis includes 59 treated subjects, with a total of 55.88 subject-years of treatment with RI-002
Measure: Number; unit: participants
Arm/Group | RI-002 Treatment
Number analyzed (Participants) | 59
participants | 36

ADVERSE EVENTS:
Time Frame: Subjects were treated with RI-002 every 3 or 4-weeks for up to 12 months, with Adverse Events reported from time of consent through the last study follow-up
Arm/Group | RI-002 Treatment
Serious Adverse Events (participants affected / at risk) | 2/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RI-002 Treatment (N=59)
Postoperative wound infection (Infections and infestations) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RI-002 Treatment (N=59)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (17)
Vomiting (Gastrointestinal disorders) | 5 (6)
Adverse drug reaction (General disorders) | 5 (8)
Fatigue (General disorders) | 8 (19)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 6 (10)
Acute sinusitis (Infections and infestations) | 11 (15)
Bronchitis (Infections and infestations) | 12 (14)
Ear infection (Infections and infestations) | 3 (4)
Gastroenteritis (Infections and infestations) | 4 (7)
Gastroenteritis viral (Infections and infestations) | 13 (16)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 13 (23)
Sinusitis (Infections and infestations) | 16 (31)
Upper respiratory tract infection (Infections and infestations) | 13 (15)
Urinary tract infection (Infections and infestations) | 6 (9)
Viral upper respiratory tract infection (Infections and infestations) | 8 (14)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Migraine (Nervous system disorders) | 8 (13)
Anxiety (Psychiatric disorders) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cough (Reproductive system and breast disorders) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication (sponsor coordinated), the Institution/PI may publish data or results from the study, if the material is reviewed by the sponsor at least 60 days prior to the proposed deadline; sponsor may remove any information considered confidential other than study data and results. If a multi-center publication is not submitted within 24 months after conclusion of the study at all sites, the Institution/PI may publish the study results following review by the Sponsor.